CLINICAL TRIAL: NCT02320591
Title: Evaluation of the Comprehensive Primary Care Initiative
Acronym: CPC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mathematica Policy Research, Inc. (Other)
Collaborators: Centers for Medicare and Medicaid Services (U.S. Federal Agency)
Responsible Party: Principal Investigator, Randy Brown, Project Director; Director of Health Services Research, Mathematica Policy Research, Inc.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HHSM-500-T0006
Record Dates: First submitted 2014-12-15; First posted 2014-12-19 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Medicare Expenditures, Quality of Care
MeSH Terms: interventions — Health Planning Technical Assistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment group (Experimental): Practices assigned to the treatment group received per member per month care management fees for each Medicare beneficiary attributed to their practice. They also received quarterly feedback reports on their patients' average Medicare expenditures and use of hospital and emergency room services. Practices also had access to regional learning faculties for technical assistance with transformation activities and to share lessons across practices.
  Interventions: Other: care management fee; Other: feedback reports; Other: technical assistance
- Comparison group (No Intervention): Within each of the 7 regions, this group is comprised of practices that were matched to the treatment practices on a wide range of baseline characteristics of the practices (including their service utilization patterns) and their patients. Comparison practices were selected from a pool of practices including those that applied to participate but were not selected, and practices serving nearby external comparison areas.

INTERVENTIONS:
Other: care management fee — for each Medicare beneficiary attributed to the practice, the practice received a monthly care management fee
  Arms: Treatment group
Other: feedback reports — Each participating practice received quarterly reports showing the practice's trend in key outcomes during the pre-intervention and intervention periods. The risk adjusted average Medicare expenditures of their patients were also shown in relation to all of the other CPC practices in their region, and to those with a similar average risk profile. Unadjusted hospitalization rates and emergency room visits were also plotted over time and compared to those of other CPC practices in the region
  Arms: Treatment group
Other: technical assistance — CPC practices could ask for technical assistance on transformation activities from a regional learning faculty (RLF). The RLF also provided seminars and other learning activities, as well as provided a forum for participating practices to share lessons they had learned.
  Arms: Treatment group

SUMMARY:
This study assesses the effects of the Centers for Medicare and Medicaid Services' Comprehensive Primary Care (CPC) initiative on physician practices, practice staff, Medicare and Medicaid costs and service utilization, quality of care, and patient outcomes. CPC provides financial resources, timely feedback on key practice outcomes, and a learning network to support practice transformation to improve quality of care and lower costs.

DETAILED DESCRIPTION:
CMS selected 7 regions (states or substate areas) to include in this study, based on commitment of other (ie, nonMedicare) payers in the area to provide financial resources to participating practices to support practice transformation to improve quality of care, reduce costs, and improve population health. 497 practices were selected from roughly 1000 applicants in the 7 regions to participate in the study. CMS pays participating practices a per member per month care management fee for each Medicare patient attributed to the practice. The practices also receive quarterly feedback on trends in their Medicare patients' use of hospital and emergency room services, Medicare expenditures, and patient outcomes from periodic surveys. Practices are expected to improve patient outcomes and lower Medicare costs per patient by using the additional resources to improve: risk-stratified care management, access and continuity of care, planned chronic and preventive care, patient and caregiver engagement, and coordination across the medical neighborhood. To remain in the study, practices must meet annual milestones for meaningful use of electronic health records and other practice features. The intervention period, which began in Fall 2012, will continue for 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Medicare beneficiary attributed to CPC practice or to a matched comparison practice. Patients are attributed to the practice from which they received the most E&M visits during the 2-year period examined.

Exclusion Criteria:

* Beneficiaries enrolled in a managed care plan.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 365076 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Medicare expenditures | 12 months
  average Medicare expenditures per month in Medicare fee-for-service

SECONDARY OUTCOMES:
number of ER visits | 12 months
  number of emergency room visits that did not result in a hospital admission
number of hospital admissions | 12 months
  number of admissions to general acute short term hospitals during the followup period
30-day hospital readmission rate | 30-days
  whether readmitted to the hospital within 30 days after discharge
hospital admission for ambulatory care sensitive condition | 12 months
  whether admitted to hospital for a condition classified as being sensitive to the quality of ambulatory care received

CONTACTS AND LOCATIONS:
Overall Officials: deborah peikes, PhD, Principal Investigator — Mathematica Policy Research; Timothy Day, MPP, Study Director — Centers for Medicare & Medicaid Services
Locations (1):
- Mathematica Policy Research, Princeton, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
not allowed; data belong to federal government (CMS)

REFERENCES:
- [Derived] Peikes DN, Swankoski K, Hoag SD, Duda N, Coopersmith J, Taylor EF, Morrisson N, Palakal M, Holland J, Day TJ, Sessums LL. The Effects of a Primary Care Transformation Initiative on Primary Care Physician Burnout and Workplace Experience. J Gen Intern Med. 2019 Jan;34(1):49-57. doi: 10.1007/s11606-018-4545-0. Epub 2018 Jul 17. PMID 30019124
- [Derived] Dale SB, Ghosh A, Peikes DN, Day TJ, Yoon FB, Taylor EF, Swankoski K, O'Malley AS, Conway PH, Rajkumar R, Press MJ, Sessums L, Brown R. Two-Year Costs and Quality in the Comprehensive Primary Care Initiative. N Engl J Med. 2016 Jun 16;374(24):2345-56. doi: 10.1056/NEJMsa1414953. Epub 2016 Apr 13. PMID 27074035